CLINICAL TRIAL: NCT06052579
Title: A Controlled Study of Articular Process Retractor Assisted- Multifidus Lateral Approach for Transforaminal Lumbar Interbody Fusion
Brief Title: Comparison Of A Novel Hand-held Retractor-Assisted Transforaminal Lumbar Interbody Fusion By The Wiltse Approach And Posterior TLIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2022-309
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Lumbar Stenosis; Spondylolisthesis
Keywords: Wiltse approach TLIF; transforaminal lumbar interbody fusion; hand-held retractors system
MeSH Terms: conditions — Constriction, Pathologic; Spondylolisthesis

STUDY DESIGN:
Intervention Model Description: This one-year prospective controlled study compared two approaches (Wiltse TLIF vs P-TLIF) for hand-held retractors-assisted TLIF was approved by the Institutional Review Board (IRB) of our hospital. Written informed consent was obtained from all study participants. 60 eligible patients were included in this study and were divided into two groups.30patientswere included in the study group and underwent Wiltse TLIF, and 30 were included in the control group and underwent P-TLIF.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): the patients included in the study group underwent Wiltse TLIF
  Interventions: Procedure: new hand-held retractor systems-assisted WiltseTLIF surgery
- control group (Active Comparator): the patients included in the control group underwent traditional posterior -TLIF
  Interventions: Procedure: new hand-held retractor systems-assisted WiltseTLIF surgery

INTERVENTIONS:
Procedure: new hand-held retractor systems-assisted WiltseTLIF surgery — patients were included in study group underwent the new hand-held retractors assisted Wiltse TLIF surgery

SUMMARY:
In recent years, hand-held retractors have been applied to assist in Wiltse approach to perform canal decompression, causing less paraspinal muscle injury and yielding better postoperative clinical outcomes than P-TLIF. However, few prospective studies have been conducted comparing the clinical and radiological outcomes between Wiltse TLIF and P-TLIF, both assisted by hand-held retractors. Therefore, further research is warranted to assess whether hand-held retractor-assisted Wiltse TLIF can yield less paraspinal muscle injury and better postoperative clinical outcomes.

DETAILED DESCRIPTION:
Study procedures How many people will participate in this study? Approximately 60 people will participate in this study conducted at the Nanfang Hospital of Southern Medical University.

Research Steps ■ Pre-study:

To determine if you are eligible to participate, the following procedures will be conducted during the screening:

Obtain your demographic and vital sign information Perform a physical examination Inquire about your medical history and concurrent medications Collect blood and urine samples for laboratory testing, imaging (X-ray, CT, MRI) If you are a fertile female, a pregnancy test will be conducted. A negative result is required for your participation in this study.

The screening results and/or results of relevant issues will help the researchers decide if you can continue with this study. If these checks indicate that you are suitable for this study, you will be informed by the researchers to proceed to visit 2 as soon as possible. If you do not meet the relevant criteria, you cannot continue to participate in this study, and the results will be communicated to you promptly.

■ Baseline Phase

If the researchers confirm that you meet the criteria for joining this trial, you will be enrolled in this study and undergo a transforaminal lumbar interbody fusion (TLIF) through either a multilevel paraspinal approach or a posterior midline approach, which will be randomly allocated (similar to drawing lots). The following procedures will be conducted during this visit:

Reconfirm your eligibility for participation Allocate you to either the multilevel paraspinal group or the posterior midline group based on randomization Conduct a physical examination and collect vital sign data Preoperative visual analog scale (VAS) score for pain, Oswestry Disability Index (ODI) score for back pain, Japanese Orthopaedic Association (JOA) score for lower back pain, and MOS 36-Item Short Form Health Survey (SF-36) quality of life score ■ Treatment Phase

During this period, the researchers will perform surgery on you based on the randomization results and assess the surgical outcomes. To ensure the accurate recording and evaluation of your condition, your cooperation is required for the following procedures:

Record postoperative drainage, time to get out of bed, discharge time, and postoperative complications Extract approximately 5ml of venous blood from you 24 hours after surgery to measure serum creatine kinase (CK) and C-reactive protein (CRP) Assess you using the VAS, ODI, JOA lower back pain score, and SF-36 quality of life score 7 days after surgery

■ Follow-up Phase

After you complete this stage of visits, it is generally considered that you have completed the entire study. The following procedures will be carried out during this period:

X-ray examination of the lumbar vertebrae in the anteroposterior and lateral views, assessment of pain, functional impairment, and quality of life score at the 3rd month after surgery X-ray and lumbar spine MRI at the 6th month after surgery, assessment of pain, functional impairment, and quality of life score X-ray and lumbar spine CT at the 1st year after surgery, assessment of pain, functional impairment, and quality of life score X-ray and lumbar spine CT at the 2nd year after surgery, assessment of pain, functional impairment, and quality of life score 3.3. What tests and assessments will be conducted in this study? After providing written informed consent, you will undergo various tests, examinations, and procedures during this study. If you have any concerns about any of these tests, please discuss them with the study doctor.

Regarding the tests and procedures for this study, we would like to provide the following information:

Medical history: The study doctor will ask you some questions to understand any current or past illnesses.

Demographic data: The study doctor will collect personal information about you, such as date of birth and ethnic background.

Physical examination: The study doctor will conduct a medical examination of your body to assess all or part of the following human body systems: head, eyes, ears, nose and throat, chest, lungs, heart, abdomen, bones, skin, neck, and nervous system.

Height and weight: Your height and weight will be measured. Vital signs: The study doctor will measure your blood pressure, heart rate, body temperature, and respiratory rate.

Blood collection: During this study, you will undergo multiple blood draws. Blood samples will be collected for the following purposes:

Preoperative blood draw: Preoperative tests (complete blood count, electrolytes, liver and kidney function, coagulation function, infection indicators), routine preoperative assessment.

Blood draw 24 hours after surgery: Approximately 5ml of venous blood will be drawn to measure serum creatine kinase (CK) and C-reactive protein (CRP).

Routine blood tests on the 3rd day after surgery: Complete blood count, ion six tests, infection two tests.

Urine samples: Routine urine tests. Pulmonary function and echocardiography if necessary. Lumbar spine anteroposterior (preoperative, 7 days after surgery, 3 months after surgery, 6 months after surgery, 1 year after surgery, 2 years after surgery), dynamic positions, oblique positions, lumbar spine MRI (preoperative and 6 months after surgery), lumbar spine CT (preoperative, 1 year after surgery, 2 years after surgery).

Questionnaire: Visual Analog Scale (VAS) score for pain, Oswestry Disability Index (ODI) score for back pain, Japanese Orthopaedic Association (JOA) score for lower back pain, and MOS 36-Item Short Form Health Survey (SF-36) quality of life score (preoperative, 7 days after surgery, 3 months after surgery, 6 months after surgery, 1 year after surgery, 2 years after surgery) How long will this study last? This clinical study will last approximately 2 years (6 visits in total). During your participation in this study, you must comply with the specified visit schedule.

You have the right to control the use and disclosure of your personal information. Where permitted by national law, you can request to view your medical information at any time. You have the right to review all information collected about you in this study and request corrections (if applicable).

New information related to the study During the study period, if there are changes in study procedures, newly discovered side effects, or significant developments that may affect your health or willingness to participate, the research team will inform you. The study doctor will notify you immediately and discuss with you whether you want to continue participating in this study. If you decide not to continue in this study, the study doctor will make arrangements for your diagnostic and therapeutic care to continue. If you choose to remain in this study, the study doctor may ask you to sign a new informed consent form.

Use of Research Results and Confidentiality of Personal Information At the end of the study, we will prepare a report and send it to the government regulatory agency. The results of this study may also be published in journals or presented at conferences, but will not contain any information that could identify you. To ensure privacy, records or samples published for research purposes will not include your name or other identifying information. Instead, your information will be identified only by a code. Only the study doctor and authorized personnel will be able to link this code to your name using a list that will be securely kept at the study center. In order to ensure that the study is conducted correctly at the study center, when necessary, the applicant, the ethics review committee, and the government regulatory authorities may review your information according to regulations. They are bound by confidentiality and will not violate your privacy.

You have the right to control the use and disclosure of your personal information. Where permitted by national law, you can request to view your medical information. You have the right to review all information collected about you in this study and request corrections (if applicable).

ELIGIBILITY:
Inclusion Criteria:

* patients underwent either one or two-level spinal fusion surgery due to lumbar stenosis, grade 1 or 2 spondylolisthesis, or lumbar disc herniation with lumbar instability and mechanical lower back pain

Exclusion Criteria:

* Patients with lumbar infection (i), spinal tumor (ii), severe osteoporosis (iii), pregnant and lactating women (iv), severe lumbar stenosis (v), and severe comorbidities (vi)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
the degree of paraspinal muscle degeneration | 6 months postoperatively
  the infiltration of fat and connective tissue are mainly manifested as enhanced signals on T2-weighted imaging

SECONDARY OUTCOMES:
the degree of paraspinal muscle degeneration | Preoperative,7 days, 3, 6, and 12 months after surgery
  concentrations of the Serum creatine kinase and C reactive-protein

CONTACTS AND LOCATIONS:
Overall Officials: Xing Shen, M.D, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Division of Spinal Surgery, Department of Orthopaedics, Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen X, Li FT, Quan Cheng Y, Zheng MH, Yao XQ, Wang HM, Ting Chen J, Jiang H. Comparison of a novel hand-held retractor-assisted transforaminal lumbar interbody fusion by the wiltse approach and posterior TLIF: a one-year prospective controlled study. BMC Musculoskelet Disord. 2024 Feb 14;25(1):142. doi: 10.1186/s12891-024-07248-w. PMID 38355528